CLINICAL TRIAL: NCT01981564
Title: Asthma Express Intervention to Bridge Emergency to Primary Care for High Risk Children With Asthma
Brief Title: Asthma Express: Bridging the Emergency to Primary Care in Underserved Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NA00078937; R01NR013486 (NIH); NCT01970085 (obsolete NCT alias)
Record Dates: First submitted 2013-10-30; First posted 2013-11-11 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Asthma
Keywords: Pediatric; Emergency department visit
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asthma Express Intervention (Experimental): Clinic visit for asthma education + nurse home visits
  Interventions: Behavioral: Asthma Express Intervention
- Standard Asthma Education Control group (Active Comparator): Standard asthma education during nurse home visits
  Interventions: Behavioral: Standard Asthma Education Control Group

INTERVENTIONS:
Behavioral: Asthma Express Intervention — Asthma Express clinic visit for asthma education + nurse home visit
  Other Names: Asthma Express
  Arms: Asthma Express Intervention
Behavioral: Standard Asthma Education Control Group — Asthma Express home nurse visits for asthma education
  Other Names: Attention Control
  Arms: Standard Asthma Education Control group

SUMMARY:
Asthma is the number one cause of pediatric emergency department (ED) visits in young minority children and is responsible for high healthcare costs. The ED is often the point of contact for many inner city children and many families view the ED as the child's primary source of asthma care. This study plans to test a new model of asthma care, Asthma Express (AEx), that includes a follow-up asthma visit in the ED for an asthma "check-up" , asthma education, a prescription for preventive asthma medications, an appointment for the child to see their pediatric provider and a home visit to assist families with environmental control methods to prevent asthma symptoms.

DETAILED DESCRIPTION:
Asthma, the leading chronic disorder in childhood, is the number one cause of pediatric emergency department (ED) visits in young children and is responsible for a substantial impact on healthcare costs. The ED is often the point of contact for low-income children and many families view the ED as their primary source of asthma care. Poor and minority children have the highest asthma morbidity, are the least likely to receive adequate preventive therapy or specialty care and more frequently exposed to environmental triggers than non-poor children. However, prior studies, including our pilot, indicate that children with frequent asthma ED visits will attend a one-time ED-based follow-up clinic for an asthma "check-up" and education. The goal of this randomized controlled trial is to test the efficacy of a multifaceted, ED + primary care provider (PCP) and home-based intervention, Asthma Express (AEx), for children with > 2 asthma ED visits or 1 hospitalization/year that provides tailored guideline based asthma care. Allergy and cotinine biomarkers, collected during the ED visit, are used to target the home environmental control component of the intervention. The AEx intervention (n=132) will be compared to an attention control (CON) group (n=132) for the specific aims: (1) to reduce asthma morbidity (increase symptom free days and nights) and decrease ED visits and hospitalizations and increase asthma control and caregiver quality of life, (2) to improve the use of appropriate preventive anti-inflammatory medication based on child pharmacy refill records and (3) to compare the economic cost and effects of this intervention. Children aged 3-12 years with > 2 asthma ED visits or 1 hospitalization within the past 12 months and a current ED visit for asthma will be recruited from the Johns Hopkins Pediatric-ED and followed for 12 months. Symptom frequency, health care utilization, caregiver quality of life and cotinine measures will be collected at baseline, 6 and 12 months and pharmacy data collected at baseline and 12 months. Data analysis includes initial cross tabulations of health outcomes by group (AEx vs. CON) and multivariate generalized linear regression models to study the effects of the AEx treatment on mean symptom free days/nights, repeat ED visits, hospitalizations and caregiver quality of life scores and anti-inflammatory medication refills. Mean total costs of ED, PCP visits, hospital days and medication costs will be compared between groups (AEx and CON) for the economic analysis. The AEx model is designed to be accessible, guideline-based, easily replicated and incorporated into ED care. If successful, this study will fill critical gaps in the ED transition to preventive care asthma interventional research.

ELIGIBILITY:
Inclusion Criteria:

* asthma diagnosis,
* age 3 to 12 years,
* two or more ED visits or one hospitalization for asthma within past 12 months, -working phone

Exclusion Criteria:

-other respiratory chronic disease such as Cystic Fibrosis or Bronchopulmonary dysplasia

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2013-04-15 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene M Butz, ScD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital Pediatric Emergency Department, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kub JE, DePriest KN, Bellin MH, Butz A, Lewis-Land C, Morphew T. Predictors of Depressive Symptoms in Caregivers of Children With Poorly Controlled Asthma: Is the Neighborhood Context Important? Fam Community Health. 2022 Jan-Mar 01;45(1):10-22. doi: 10.1097/FCH.0000000000000313. PMID 34783687
- [Derived] Margolis RHF, Dababnah S, Sacco P, Jones-Harden B, Bollinger ME, Butz A, Bellin MH. The Effects of Caregiver Social Support and Depressive Symptoms on Child Medication Adherence and Asthma Control. J Racial Ethn Health Disparities. 2022 Aug;9(4):1234-1242. doi: 10.1007/s40615-021-01065-w. Epub 2021 May 26. PMID 34041705
- [Derived] Margolis RHF, Bellin MH, Bookman JRM, Collins KS, Bollinger ME, Lewis-Land C, Butz AM. Fostering Effective Asthma Self-Management Transfer in High-Risk Children: Gaps and Opportunities for Family Engagement. J Pediatr Health Care. 2019 Nov-Dec;33(6):684-693. doi: 10.1016/j.pedhc.2019.05.004. Epub 2019 Jun 26. PMID 31253454
- [Derived] Bollinger ME, Butz A, Tsoukleris M, Lewis-Land C, Mudd S, Morphew T. Characteristics of inner-city children with life-threatening asthma. Ann Allergy Asthma Immunol. 2019 Apr;122(4):381-386. doi: 10.1016/j.anai.2019.02.002. Epub 2019 Feb 10. PMID 30742915
- [Derived] Butz AM, Tsoukleris M, Elizabeth Bollinger M, Jassal M, Bellin MH, Kub J, Mudd S, Ogborn CJ, Lewis-Land C, Thompson RE. Association between second hand smoke (SHS) exposure and caregiver stress in children with poorly controlled asthma. J Asthma. 2019 Sep;56(9):915-926. doi: 10.1080/02770903.2018.1509989. Epub 2018 Oct 11. PMID 30307351
- [Derived] Bellin MH, Newsome A, Lewis-Land C, Kub J, Mudd SS, Margolis R, Butz AM. Improving Care of Inner-City Children with Poorly Controlled Asthma: What Mothers Want You to Know. J Pediatr Health Care. 2018 Jul-Aug;32(4):387-398. doi: 10.1016/j.pedhc.2017.12.009. Epub 2018 Mar 12. PMID 29540280
- [Derived] Butz AM, Bellin M, Tsoukleris M, Mudd SS, Kub J, Ogborn J, Morphew T, Lewis-Land C, Bollinger ME. Very Poorly Controlled Asthma in Urban Minority Children: Lessons Learned. J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):844-852. doi: 10.1016/j.jaip.2017.08.007. Epub 2017 Sep 22. PMID 28958744
- [Derived] Butz A, Morphew T, Lewis-Land C, Kub J, Bellin M, Ogborn J, Mudd SS, Bollinger ME, Tsoukleris M. Factors associated with poor controller medication use in children with high asthma emergency department use. Ann Allergy Asthma Immunol. 2017 Apr;118(4):419-426. doi: 10.1016/j.anai.2017.01.007. Epub 2017 Feb 21. PMID 28254203
- [Derived] Bellin MH, Newsome A, Land C, Kub J, Mudd SS, Bollinger ME, Butz AM. Asthma Home Management in the Inner-City: What can the Children Teach us? J Pediatr Health Care. 2017 May-Jun;31(3):362-371. doi: 10.1016/j.pedhc.2016.11.002. Epub 2016 Dec 9. PMID 27955875
- [Derived] Bellin MH, Land C, Newsome A, Kub J, Mudd SS, Bollinger ME, Butz AM. Caregiver perception of asthma management of children in the context of poverty. J Asthma. 2017 Mar;54(2):162-172. doi: 10.1080/02770903.2016.1198375. Epub 2016 Jun 15. PMID 27304455
- [Derived] Butz AM, Ogborn J, Mudd S, Ballreich J, Tsoukleris M, Kub J, Bellin M, Bollinger ME. Factors associated with high short-acting beta2-agonist use in urban children with asthma. Ann Allergy Asthma Immunol. 2015 May;114(5):385-92. doi: 10.1016/j.anai.2015.03.002. Epub 2015 Mar 31. PMID 25840499

RESULTS

PARTICIPANT FLOW:
Groups:
- Asthma Express Intervention: Clinic visit for asthma education + nurse home visits
  Asthma Express Intervention: Asthma Express clinic visit for asthma education + nurse home visit
  Asthma Express Control Arm: Asthma Express home nurse visits for asthma education
- Standard ASthma Education Control Group: STandard asthma education delivered in home by nurse
  Asthma Express Intervention: Asthma Express clinic visit for asthma education + nurse home visit
  Asthma Express Control Arm: Asthma Express home nurse visits for asthma education
Period: Overall Study
Arm/Group | Asthma Express Intervention | Standard ASthma Education Control Group
Started | 107 | 115
Completed | 98 | 106
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthma Express Intervention | Standard ASthma Education Control Group | Total
Number analyzed (Participants) | 107 | 115 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 107 | 115 | 222
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (2.7) | 6.5 (2.6) | 6.3 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 35 | 80
  Male | 62 | 80 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 103 | 112 | 215
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 101 | 107 | 208
  White | 4 | 3 | 7
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 107 | 115 | 222
Symptoms days past 14 days [Mean (Standard Deviation); unit: symptom days] | 5.55 (4.6) | 6.17 (4.9) | 5.88 (4.8)
Emergency Department visits over past 3 months [Mean (Standard Deviation); unit: Number of ED visits over past 3 months] — Population: 3 caregivers did not report number of ED visits over past 3 months at the baseline survey.
  Number of ED visits over past 3 months
    number analyzed (Participants) | 105 | 114 | 219
    (all) | 1.02 (1.1) | 1.48 (1.6) | 1.26 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Symptom Days
Description: Symptom days for asthma during past 14 days
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: symptom days over past 14 days
Arm/Group | Asthma Express Intervention | Standard ASthma Education Control Group
Number analyzed (Participants) | 98 | 106
symptom days over past 14 days | 6.24 (5.7) | 4.82 (5.1)
Statistical Analysis 1: Comparison: Asthma Express Intervention; ANOVA F=3.55, df=1, p=0.06; Test type: Superiority; p = 0.06, ANOVA

2. Secondary Outcome: Emergency Department (ED) Visits for Asthma
Description: Number of emergency department visits for asthma in the past 3 months
Time Frame: 3 months
Population: No data for one participant in the control group for this outcome
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Asthma Express Intervention | Standard Asthma Education Control Group
Number analyzed (Participants) | 98 | 105
visits | 0.64 (2.26) | 0.62 (1.02)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Asthma Express Intervention | Standard ASthma Education Control Group
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/106
Other Adverse Events (participants affected / at risk) | 0/98 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT01981564/Prot_SAP_000.pdf